CLINICAL TRIAL: NCT06681896
Title: Microvascular Coronary Rehabilitation For Improving Treatment - Feasibility Study
Acronym: MICROFIT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Royal United Hospitals Bath NHS Foundation Trust (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 340782; TRP23-100023 (Other Grant/Funding Number: Heart Research UK); 64259 (Other Grant/Funding Number: NIHR Research Delivery Network)
Record Dates: First submitted 2024-11-05; First posted 2024-11-12 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2024-11

CONDITIONS: Microvascular Coronary Dysfunction; Microvascular Angina; Coronary Microvascular Dysfunction (CMD)
Keywords: coronary microvascular dysfunction; HIIT; high intensity interval exercise training; exercise training; dietary rehabilitation; lifestyle advice; microvascular angina
MeSH Terms: conditions — Microvascular Angina | interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MICROFIT + Usual Care (Experimental): MICROFIT intervention will be delivered in addition to Usual Care arm clinical review and advice. MICROFIT is a 24-week long personalized one-on-one exercise and dietary education intervention, along with home exercise guided by personal trainers. Exercise intervention includes High Intensity Interval Training (HIIT) and dietary advice focuses on incorporation of a Mediterranean-type diet.
  Interventions: Other: MICROFIT - personalised high intensity interval training exercise rehabilitation and dietary advice
- Usual Care (No Intervention): All patients will be reviewed clinically by a cardiologist. They will address cardiovascular risk factors and prescribe any therapies as indicated by current medical guidelines, for example statin or ACE inhibitors. The Cardiologist will also provide routine, verbal one-off lifestyle advice in line with NICE guidance, recommending 150 minutes of moderate exercise per week, encouraging a healthy, balanced diet, weight loss, reducing alcohol consumption and smoking cessation where necessary.

INTERVENTIONS:
Other: MICROFIT - personalised high intensity interval training exercise rehabilitation and dietary advice — MICROFIT is a 24-week long personalized one-on-one exercise and dietary education intervention, along with home exercise guided by personal trainers. Exercise intervention includes High Intensity Interval Training (HIIT) and dietary advice focuses on incorporation of a Mediterranean-type diet.
  Phase 1 - Induction (8 weeks) Exercise: Twice-weekly 1-hour personal trainer (PT) supervised exercise sessions. 45 minute homework exercise session once a week.
  Diet: 1-hour educational session with a dietician, followed by two 30-minute follow up sessions.
  Phase 2 - Consolidation (10 weeks) Exercise: Once weekly 1 hour PT sessions, two 45 minute homework sessions once a week.
  Diet: 30-minute sessions every 5 weeks.
  Phase 3 - Maintenance (6 weeks) Exercise: Supervised 1 hour PT sessions once every 3 weeks, 45-minute homework sessions three times a week.
  Diet: one final 30 minute session after week 3.
  Arms: MICROFIT + Usual Care

SUMMARY:
The goal of this clinical trial is to assess the feasibility of undertaking a randomized controlled trial assessing the impact of a personalised, intense cardiac rehabilitation programme involving high intensity interval exercise (HIIT) and dietary advice (termed MICROFIT) on symptom burden in patients with microvascular coronary dysfunction.

The main questions it aims to answer are:

1. Feasibility of undertaking randomised controlled trial of MICROFIT in patients with coronary microvascular dysfunction (recruitment rates, retention and adherence, acceptability of MICROFIT and participants' and practitioners' experiences of trial participation)
2. Preliminary data on the effect that MICROFIT has on angina symptoms in patients with microvascular coronary dysfunction, as measured by Seattle Angina Questionnaire
3. Preliminary data on the fidelity and clinical efficacy of MICROFIT

Participants will be randomized to either MICROFIT + Usual Care, or Usual Care group.

Participants in both arms of the trial will:

* Undergo a series of investigations, including cardiopulmonary exercise test (CPET), dual xray absorptiometry (DEXA), echocardiogram, cardiac MRI scan, blood tests, at the start of the trial and again after 6 months
* Measure their living activity by using an activity tracker (GeneActiv) as well as a photographic diet diary for a week at the start of the trial and again after 6 months
* Complete a series of questionnaires to assess angina symptom burden, mental health and quality of life, at the start of the trial and again after 6 months.

Participants in the intervention arm of the study will:

1. Undergo MICROFIT intervention. MICROFIT includes a combination of exercise and diet management sessions over 24 weeks. It involves:

   * 1:1 high-intensity interval training ('HIIT') sessions with a personal trainer and guidance on exercise sessions to be performed at home
   * 1:1 sessions with a dietician to support them with improvements in diet.
2. Visit clinic on two additional occassions during the trial to discuss their progress with a cardiologist
3. Undergo an interview at the end of the study to discuss their experiences of participation in the study
4. Receive a debrief on their investigation results and progress made at the end of their study

Participants in the Usual Care arm of the study will:

1. Receive standard Usual Care advice regarding lifestyle changes and targeted medical therapy offered to patients with coronary microvascular dysfunction.
2. Receive a debrief on their investigation results and progress made at the end of their study
3. Undergo a 'taster' session with the personal trainer to discover what the intervention involves.

DETAILED DESCRIPTION:
The investigators hypothesise that an intensified and personalised healthcare delivered lifestyle intervention (MICROFIT) will improve anginal symptoms in patients with microvascular coronary dysfunction. As a first step to a multi-centre randomised controlled trial (RCT) to establish efficacy, this feasibility study will test the components and acceptability of the intervention, alongside preliminary data on change in anginal symptoms to guide the powering of the subsequent RCT.

Participants:

The investigators aim to recruit 40 participants (men and women) with confirmed coronary microvascular dysfunction identified via existing clinical pathways (following an invasive coronary angiography study resulting in a diagnosis of microvascular angina) at two study sites, the Royal United Hospitals Bath NHS Foundation Trust (RUH) and University Hospitals Bristol and Weston NHS Foundation Trust(UHBW). Invasive coronary angiography with a microvascular study is a gold standard assessment for microvascular dysfunction nationwide and thus would be transferrable to all sites in the proposed subsequent multicentre randomised controlled trial.

A named cardiologist at each site who will be a member of the research team will undertake the screening. Potential participants will be approached on the day of their attendance for microvascular dysfunction testing following the procedure, once microvascular dysfunction has been confirmed (as per inclusion criteria), or during a routine follow up appointment as part of usual care relating to the diagnosis of coronary microvascular disease. Potential participants will be informed of the experimental protocol both verbally and in writing before providing informed consent. The study will be conducted in accordance with the Declaration of Helsinki. Participants will be block randomised 1:1 using a web-based platform (Sealed Envelope: https://www.sealedenvelope.com/). Participants will be randomised to either usual care (control arm) or MICROFIT with usual care, in permuted blocks of four and stratified for sex. The control arm contributes to a robust assessment of feasibility (e.g. consent and attrition rates) and a comparator for the preliminary data on anginal symptom burden change.

TRIAL ARMS:

Usual care (control arm):

All patients will be reviewed clinically by the Cardiologist performing the initial assessment. The cardiologist will address cardiovascular risk factors and prescribe any therapies, for example aspirin or statin therapy, as indicated by NICE guidelines. The Cardiologist will have over-arching responsibility for patients involved in the study, however, each patient's General Practitioner will be provided with a study information sheet and encouraged to adjust medications as needed according to national guidelines (e.g. for diabetic or hypertension management if these improve whilst participating in the study). The Cardiologist will also provide routine, verbal one-off lifestyle advice in line with NICE guidance, recommending 150 minutes of moderate exercise per week, encouraging a healthy, balanced diet, weight loss, reducing alcohol consumption and smoking cessation where necessary. The participants in the usual care arm will undergo the same assessments at baseline and at 24 weeks as the MICROFIT + Usual care arm, following which they will be offered a taster session with the personal trainer as well as information booklet regarding dietary advice offered to the participants in the MICROFIT + Usual Care arm.

MICROFIT + usual care (intervention arm):

MICROFIT is a lifestyle intervention designed to enable and support successful behavioural change with a predominant focus on exercise and diet. There is a focus on 1-on-1 delivery, higher intensity exercise, and updated dietary advice that aligns with the latest evidence-base for both microvascular dysfunction and broader cardiovascular disease. The programme will be explicitly introduced to each participant by the Cardiologist to ensure that the programme is presented as a meaningful intervention that can improve health outcomes. From the patient perspective, the Cardiologist will be seen as leading a multidisciplinary team, including exercise trainers and nutritional advisors, who are collectively working to improve the patient's microvascular function, measured both in terms of symptoms as well as objectively through stress perfusion MRI. The Cardiologist will introduce the concepts involved in the nutritional advice to the participant in the introductory session, provide advice and oversight to both the nutritional and exercise trainers throughout, and conduct further clinical reviews at the end of each intervention phase.

MICROFIT has three phases: (1) induction, (2) consolidation and (3) maintenance. Below the structure of different phases of MICROFIT trial delivery is summarised. The exercise and dietary components are further explained in the next section.

Phase 1 - Induction (8 weeks) Exercise: Twice-weekly 1-hour exercise trainer supervised exercise sessions (described below), with once-weekly sessions of prescribed moderate-intensity "homework". Weekly body metrics (BP, HR, BMI) will enable goal-setting and feedback to encourage adherence.

Diet: Baseline 1-hour educational session with a dietician, followed by two 30 minute follow up sessions. These will be delivered virtually or face to face.

Phase 2 - Consolidation (10 weeks) Exercise: Reduced supervised session frequency to once-weekly, with two sessions of prescribed moderate-intensity homework/week. Body metrics 2-weekly.

Diet: 2x 30-minute "touch-base" sessions every 5 weeks, providing ongoing behavioural support of self-monitoring and goals.

Phase 3 - Maintenance (6 weeks) Exercise: Supervised sessions reduced to one every 3 weeks, with three times/week prescribed sessions of homework (now higher-intensity aerobic exercise). Body metrics assessed at penultimate visit.

Diet: A 30-minute "touch-base" session responding to changes in behaviour, where necessary.

Below each component of the MICROFIT intervention is explained.

Exercise Component:

(i)Supervised Sessions: Experienced exercise trainers will lead supervised 1:1 exercise sessions incorporating HIIT based on the Norwegian4x4 model for CAD patients. At the start of each supervised exercise session, participants will be asked about any change in symptoms or medications and have blood pressure and heart rate measured. Participants will be taught the Borg Rating of Perceived Exertion (RPE; 6-20). The acceptable maximal heart rate will be calculated upon patient's age baseline CPET results, adjusted as recommended for patients taking beta-blockers. The first session will consist of a graduated, lead-in of moderate intensity exercise prior to commencement of HIIT in subsequent sessions. Supervised sessions will use a cardiovascular exercise (e.g. static bike or treadmill) and HIIT sessions will comprise a 3-minute warm-up; four 4- minute high-intensity intervals at RPE 15 (hard), finishing at RPE 17-18 (very hard); 3 minutes of active recovery at RPE 11-13 (somewhat hard) between each interval; and conclude with 5-minute recovery as is advised for patients with cardiovascular disease. Trainers will help maintain target intensity and monitor participants throughout for concerning symptoms. To enable this and mitigate risk, all trainers will be required to complete a MICROFIT training course that will incorporate symptom supervision, basic life support and defibrillator training. All exercise facilities will have a defibrillator on site. In addition, given the benefits of resistance exercise, especially for blood pressure control, the sessions will conclude with twenty minutes of resistance training. The exercise trainer will feedback power data to participants as they work through the programme to highlight visible progress being achieved.

(ii) Homework Sessions: To enhance the weekly workload achieved and support long-term behaviour change, participants will be prescribed "homework" exercise sessions. This will comprise moderate-intensity aerobic exercise for 45-minutes in induction and consolidation phases (e.g., brisk walking), and increase to higher-intensity exercise (e.g., hill walking or jogging) in the maintenance phase. A once weekly resistance exercise session using workouts learnt in the supervised session during phases 1 and 2 will be added in phase 3. Participants will be provided with written guidance on effort levels, how to monitor their symptoms, and a HR monitor (MyZone) to support self-directed exercise intensity, ensuring their intensity is at the appropriate level. These data will be reviewed at supervised exercise sessions by personal trainers to evaluate progress and provide support and kept for subsequent analysis.

Dietary Component:

Patients will complete pre-session combined photographic/written diet diaries (retained by the research team for dietary analysis). Recognising that there is no "one-size-fits-all" pattern, the nutritional advisor will work with the patient to identify residual barriers to dietary change and potential solutions. The photographic diet diary will help highlight incremental areas for improvement in a straightforward manner. Where indicated, the dietician will also continue to highlight the importance of smoking cessation during sessions. The principles and guiding framework for the dietary advice will be:

* Adoption of the Mediterranean-style diet in everyday diet
* Reduced carbohydrate intake, focusing on avoidance of starch-based vegetables and refined grains
* Reduced added sugars, using diet diaries to highlight "hidden sugars"
* Drinking water (no smoothies, diet drinks, juices), unsweetened tea/coffee and alcohol in moderation
* Avoidance of ultra-processed foods, e.g., highly-processed meat
* Avoidance of "low-fat" products, in favour of natural, whole foods with unsaturated and/or mono-saturated fats
* Increased dietary fibre
* Focus on dietary patterns, including advice to eat at regular mealtimes and portion control rather than "calorie counting", alongside snack reduction and identifying healthy alternatives. The participants will be offered an information booklet regarding dietary advice which they will be able to refer to throughout the course of the study.

TRIAL ASSESSMENTS:

The trial comprises of five assessment episodes:

1. baseline assessment prior to participant randomisation, part of which is undertaken for convenience at the sametime as screening and consent visit
2. in-study assessment at 8 weeks
3. in-study assessment at 18 weeks
4. end of study assessment at 24 weeks
5. follow up qualitative interview 1 month after participant trial completion.

Participants in the intervention arm will undertake assessments 1-5, whereas participants in the usual care arm will attend assessments 1 and 4 only.

Assessments 1 and 4 will require attendance at RUH or UHBW (depending on participant's recruiting hospital), University of Bath and St Joseph's Hospital, Newport. Assessments 2 and 3 will require attendance at RUH or UHBW only. Assessment 5 will be undertaken face to face or virtually according to participant preference.

In order to minimise travel and appointment burden for patients, part of baseline assessment 1 will take place at the same time as screening visit. During this visit some of the baseline clinical investigations will be undertaken (including blood tests (HbA1c, lipid profile, inflammatory markers),ECG, echocardiography (if not performed within last 6 months), body anthropometrics (height, weight, waist and hip circumference), clinic BP measurement and patient questionnaires (Seattle Angina Questionnaire, Hospital Anxiety and Depression Scale and EuroQol-5D-5L questionnaire for quality of life). The patients will also be issued blood pressure monitor for 7-day home BP monitoring and wearable activity device (GeneACTIV), alongside instructions for diet diary to be undertaken at home. The participant will also be made an appointment to attend Cardiac MRI at St Joseph's Hospital and CPET (cardiopulmonary exercise test to assess fitness levels) and body composition testing (DEXA) at University of Bath. This concludes baseline Assessment 1. Assessment 4, concluding the trial, will follow the same structure.

Assessments 2 and 3 will take place solely with participants in the intervention arm of the trial. These visits will take place at RUH or UHBW and will comprise clinical review, blood tests, body anthropometrics and clinic BP.

Assessment 5 will take place face to face or virtually and will comprise of a qualitative interview on participant experience in the trial. All 20 intervention participants will be invited for a 30 - 40-minute interview upon completion to capture all ranges of experiences of participation in the trial. Interviews will seek feedback on trial participation, including barriers and facilitators to trial procedures, exercise adherence, and explore any unanticipated effects of taking part. Encrypted interviews will be recorded, transcribed verbatim and analysed using both narrative and thematic analysis.

In-depth (30 - 40 minute) interviews will be conducted with all practitioners involved in delivering MICROFIT to identify areas that need to be adapted or changed to implement the intervention in a future trial (or rollout). Specifically, this will include their experience of delivering and supporting MICROFIT, the quality of the training resources, and how participation affected their other work and relationships with patients.

MICROFIT adherence measurement:

Adherence to MICROFIT will comprise of attendance at supervised exercise and nutritional sessions, and participation in home unsupervised sessions.

A summary of the assessments at each time points is shown in Trial Flowchart within trial Protocol.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18
* Angina or angina equivalent symptoms
* Unobstructed coronary arteries at the time of coronary angiogram. This will be defined as plaque causing <40% epicardial vessel stenosis or 40-90% with a fractional flow reserve (FFR) ≥0.8
* Evidence of microvascular dysfunction on ICA (CFR <2.5 and/or AchFR <1.5)

Exclusion Criteria:

* New York Heart Association class III/IV heart failure
* Severe left ventricular impairment (ejection fraction≤35%)
* Severe heart valve disease
* Significant cardiomyopathy (as assessed by a cardiologist)
* Severe hypertension (defined as blood pressure >180/120mmHg (despite three anti-hypertensive agents)
* Uncontrolled arrhythmia
* A history of aortic dissection, recent (<6 months) acute pulmonary embolus, deep vein thrombosis, stroke or transient ischaemic attack, severe autonomic or peripheral neuropathy, acute systemic illness or fever, severe acute or chronic renal failure, severe pulmonary fibrosis or interstitial lung disease (in line with other trials investigating HIIT exercise)
* Pregnancy or breastfeeding (at any point during the study. Patients becoming pregnant during the study will be asked to withdraw due to additional radiation exposure and risks from HIIT)
* Physical inability to participate in exercise
* Significant claustrophobia or metallic implants which would limit MRI imaging
* Intolerance to regadenoson testing (high degree atrioventricular block, severe asthma or airways disease)
* Current participation in another intervention-based trial
* Inability to fully understand the verbal and written descriptions of the study and instructions provided during the study duration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-11-12 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Establish recruitment rate | Week 0
  A key feasibility outcome for a potential future randomised controlled trial will be to establish recruitment rates: defined as the proportion of eligible patients who accept the invitation to participate in the study.
Establish retention rate | Week 24
  A key feasibility outcome for a potential future randomised controlled trial will be to examine retention: defined as the proportion of recruited participants who complete the study.
Establish adherence | Week 24
  A key feasibility outcome for a potential future randomised controlled trial will be to examine adherence: defined as, for participants in the intervention arm, the proportion of offered sessions completed.
Assess acceptability of the intervention | Week 24
  A key feasibility outcome for a potential future randomised controlled trial will be to examine the acceptability of the intervention (MICROFIT) to participants and clinicians. This will be assessed qualitatively by an end of study interview.
Assess acceptability of the study design | Week 24
  A key feasibility outcome for a potential future randomised controlled trial will be to examine the acceptability of the study design. This will be assessed qualitatively by an end of study interview.

SECONDARY OUTCOMES:
Change in anginal symptom burden | Week 24
  Data on anginal symptom burden as measured by the 7-item Seattle Angina Questionnaire (SAQ-7) [0-100, 0=worst health, 100=full health] will be collected to guide power calculations for large scale RCT in the future, where it would be the primary outcome.
Change in myocardial perfusion with quantitative stress MRI | Week 24
  An assessment of change in myocardial perfusion reserve [ratio of myocardial blood flow at hyperaemia/myocardial blood flow at rest] utilising quantitative stress perfusion cardiac MRI.
Change in myocardial oxygenation | 24 weeks
  Qualitative and quantitative assessment of change in myocardial oxygenation utilising Oxygenation-Sensitive Cardiac MRI
Change in cardiorespiratory fitness | 24 weeks
  Serial cardiopulmonary exercise tests will provide a measurement of maximum rate of oxygen consumption attainable during physical exertion (VO2 peak), reported in mL/kg/min.
Change in blood pressure control | 24 weeks
  Participants will undertake 7-day blood pressure monitoring at home, the results of which will be averaged [mmHg]
Change in body fat composition | 24 weeks
  Changes in body fat composition will be assessed with dual-energy X-ray absorptiometry (DEXA).
Change in body anthropometrics (Body Mass Index - BMI) | 24 weeks
  Change in body mass index (BMI) will be reported using aggregated height (metres) and weight (kilograms) to arrive at one reported value (kg/m^2).
Change in anthropometrics - waist circumference | 24 weeks
  Change in abdominal waist circumference (centimetres) will be reported.
Change in glucose control, measured with the glycated haemoglobin test (HbA1c) | 24 weeks
  Serial blood sampling for HbA1c (mmol/mol)
Change in serum lipid levels | 24 weeks
  Serial blood samples will be taken to assess serum lipid profile (total cholesterol, [mmol/L], LDL cholesterol [mmol/L], HDL cholesterol [mmol/L], triglycerides [mmol/L])
Change in serum inflammatory markers | 24 weeks
  Serial blood testing to assess C-reactive protein (CRP) (mg/L)
Change in left ventricular ejection fraction, measured on echocardiography | 24 weeks
  An assessment of cardiac systolic function, defined by left ventricular ejection fraction, will be performed using echocardiography.
Change in left ventricular strain assessed on echocardiography | 24 weeks
  An assessment of cardiac systolic function, defined by left ventricular strain, will be performed using echocardiography.
Change in left ventricular filling pressure measured on echocardiography | 24 wees
  An assessment of cardiac diastolic function, with echocardiography measure of left ventricular filling pressure.
Change in left atrial strain, measured on echocardiography | 24 weeks
  An assessment of left atrial strain, a marker of diastolic dysfunction, will be performed using echocardiography.
Change in self-perceived mental health, assessed with the Hospital Anxiety and Depression Scale (HADS) | 24 weeks
  Hospital Anxiety and Depression Scale (HADS). Scores range from 0 to 21 with higher scores reflecting a higher degree of anxiety and/or depression.
Change in patient reported health-related quality-of-life, measured with the EuroQol Group (EuroQol) EQ-5D-5L questionnaire | 24 weeks
  Patient reported health-related quality-of-life will be recorded using the EuroQol EQ-5D-5L questionnaire.
Evaluate data collection procedures | Week 24
  To confirm that all data collection procedures (clinical, intervention and health economic data points) are achievable. This will be assessed as a percentage of the total number data-points we attempt to collect.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Khavandi, Principal Investigator — Royal United Hospitals Bath NHS Foundation Trust
Locations (2):
- United Kingdom (2):
  - Royal United Hospitals Bath NHS Foundation Trust, Bath
  - University Hospitals Bristol and Weston NHS Foundation Trust, Bristol

IPD SHARING:
Plan to Share IPD: Yes
All IPD collected as part of trial
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Beginning 1 month after publication of results and ending 5 years after
Access Criteria: Requests for data sharing will be reviewed on an individual basis upon request to the research team.